CLINICAL TRIAL: NCT01314638
Title: Etude de l'adhérence et Des Effets Des Ateliers "équilibre Siel Bleu" Sur la Marche, la Cognition, l'Autonomie et l'indépendance Des Sujets Atteints d'Une Maladie d'Alzheimer, et Sur le Fardeau de l'Aidant Principal
Brief Title: Study of Adherence and Effects of Balance Exercices (SIEL BLEU Associatio)
Acronym: SIELBLEU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: ANNWEILER Cédric ; MD, University Hospital, Angers
Other Study IDs: 2009-A01148-49
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Gait Apraxia; Alzheimer Disease; Impaired Cognition
MeSH Terms: conditions — Gait Apraxia; Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single group: Single group, Identical investigations for all subjects
  Interventions: Other: Workshop balances

INTERVENTIONS:
Other: Workshop balances — one workshop per week for 20 weeks. Evaluation before and after.
  Other Names: Workshop balances (SIEL BLEU Association)

SUMMARY:
The purpose of this study is to measure the adherence to "Siel bleu" balance exercises in patients with Alzheimer's disease, while taking into account the disease stages.

DETAILED DESCRIPTION:
The practice of physical activity, more specifically postural balance exercises, is an intervention that improves gait performance in the elderly. Among patients with Alzheimer's disease, it seems that physical exercice also improves cognitive performance, reduces the loss of autonomy and independence in activities of daily living. All these effects may reduce the caregiver burden.

Despite several initiatives in France, no study has been carried out to test the adherence to postural balance exercises and to examine the benefits on older AD patients and their caregiver.

The main objective of this study is to measure the adherence to "Siel bleu" balance exercises in patients with Alzheimer's disease, while taking into account the disease stages.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alzheimer's disease (AD) (DSM-IV/NINCDS-ADRDA criteria)
* Age ≥ 65 years old
* Mild AD (Mini-Mental State Examination score between 21 and 25), moderate AD (Mini-Mental State Examination score between 10 and 20) and severe AD (Mini-Mental State Examination score between 3 and 9)
* Able to walk without any aid on 15 meters.
* Near visual acuity ≥ 2
* Absence of severe depression (score of the 15-item Geriatric Depression Scale ≤ 10)
* Written consent form to participate in the study (or trustworthy person or legal representative for severe AD)
* Being affiliated to a social security regime

Exclusion Criteria:

* Musculoskeletal disorders not related to Alzheimer's disease
* Near visual acuity < 2
* History of cerebrovascular accident or other cerebro-spinal pathology
* Poor workmanship of the written or oral French language
* Refusal to be informed on possible hanging bare anomaly during study
* Score of Mini-Mental State Examination < 3
* Presence of severe depression (score of the 15-item Geriatric Depression scale > 10)
* Use of walking aid
* Subject suffering from pre-existing impellent disturbances
* Refusal to participate (or trustworthy person or legal representative)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All patients of Angers University Memory Center, with respect to the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to "Siel Bleu" balance exercices | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Cedric ANNWEILER, MD, Principal Investigator — University Memory Centre ANGERS
Locations (1):
- Angers University Hospital, Angers, France